CLINICAL TRIAL: NCT02793687
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Efficacy and Safety of Mexidol® in Long-term Sequential Treatment of Patients in the Acute and Early Recovery Periods of Hemispheric Ischemic Stroke (EPICA)
Brief Title: Study of Efficacy and Safety of MEXIDOL® in Ischemic Stroke Therapy
Acronym: EPICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPICA; 2013-08-11 (Other: Ministry of Health, Russian Federation)
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Neuroprotective Agents; Nootropic Agents; Antioxidants; Randomized Controlled Trials as Topic; Recovery of Function; Mexidol; Ethylmethylhydroxypyridine Succinate; Brain Ischemia; Acute Stroke; Acute Cerebrovascular Accident; Cerebral Stroke; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mexidol® (Experimental): Participants received Mexidol® solution IV 500 mg daily for 10 days, then Mexidol 125 mg orally 1 tablet 3 times a day for 8 weeks.
  Interventions: Drug: Mexidol
- Placebo (Placebo Comparator): Participants received Mexidol Placebo matching Mexidol solution IV 500 mg daily for 10 days, then Mexidol 125 mg orally 1 tablet 3 times a day for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mexidol — 50 mg/ml IV solution, 125 mg tablet
  Other Names: Ethylmethylhydroxypyridine Succinate
  Arms: Mexidol®
Other: Placebo — Placebo IV solution, Placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long-term sequential therapy with Mexidol® in long-term sequential treatment of patients in the acute and early recovery periods of hemispheric ischemic stroke (IS). This is superiority trial that investigates whether Mexidol® better than placebo.

DETAILED DESCRIPTION:
In the course of a clinical study involving patients, the efficacy and safety of prolonged sequential therapy with Mexidol® (solution for intravenous and intramuscular administration / coated tablets) were evaluated compared to placebo in patients with hemispheric ischemic stroke during the acute and early recovery periods. The use of Mexidol® (solution for intravenous and intramuscular administration / coated tablets) and placebo (solution for intravenous and intramuscular administration / coated tablets) was conducted against the background of standard baseline therapy.

Throughout the study, both the investigational drug Mexidol® and the placebo, used alongside baseline therapy, were tolerated satisfactorily. In this clinical study, 37 cases of adverse events (AEs) not meeting the criteria for severity were recorded in 28 patients, along with 4 AEs that were categorized as serious adverse events (SAEs) in 4 patients. Most of the registered AEs required appropriate corrective therapy but did not necessitate other medical interventions and resolved by the end of the patient's participation in the study. According to the researchers, in the majority of recorded AEs, the relationship with the investigational drugs was determined to be absent (no relationship).

When comparing the frequency of registration of both individual AEs and SAEs, no statistically significant differences (p < 0.05) were found in the frequency of AEs/SAEs in patients after taking the investigational drug (Mexidol®) and the comparison drug (placebo). According to the conducted clinical study, the safety profile of Mexidol® remained unchanged and favorable. No new safety signals were recorded during the course of the study.

The primary endpoint is the results of testing using the modified Rankin Scale (mRS) at the end of the therapy course (in both the investigational and control groups). In the overall population of patients included in the efficacy analysis, positive dynamics were observed in both the Mexidol® group and the placebo group (p < 0.001): a decrease in the mean scores on the scale throughout the study; a statistically significant difference was also identified between the mean scores on the mRS at visit 5 compared to baseline values (visit 1) in both groups. Additionally, at visit 5, a statistically significant difference was observed between the treatment groups (p = 0.04) regarding the total scores on the modified Rankin Scale: the average score for the Mexidol® group was 1.098 points, while for the placebo group, it was 1.46 points. No statistically significant differences between the groups were found at other visits. The assessment of the change in mRS score from baseline (visit 1) to the end of therapy (visit 5) showed statistically significant differences (p = 0.04) between the treatment groups: in the Mexidol® group, the value was 1.098; in the placebo group, it was 1.460.

Thus, Mexidol® demonstrated greater efficacy compared to placebo when used alongside baseline therapy in patients with hemispheric ischemic stroke during the acute and early recovery period based on the primary efficacy criterion, which is the results of testing using the modified Rankin Scale (mRS) at the end of the therapy course.

Furthermore, the study demonstrated the efficacy of Mexidol® therapy concerning several secondary efficacy endpoints. Mexidol® showed greater efficacy in treating hemispheric ischemic stroke compared to placebo when using the specialized scale for this condition-the NIHSS (National Institutes of Health Stroke Scale). In testing using the Beck Depression Inventory (BDI), the efficacy of Mexidol® regarding cognitive disorders in patients who suffered strokes with concurrent diabetes was also identified.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of first-ever hemispheric ischemic stroke (codes ICD-10: I63.0 - I63.9).
2. Age 18-80 years
3. The ability to understand the purpose of research, risks associated with the research intervention, obligations and consequences of research participation and their right of withdrawing consent any time during the study.
4. The time from onset of a stroke <72 hours.
5. The Modified Rankin Scale (mRS) score ≥3.
6. The National Institutes of Health Stroke Scale (NIHSS) score from 5 to 15 points.
7. The Beck Depression Inventory (BDI) score <19 points.
8. The written informed consent form (ICF) is signed and personally dated by the participant or by an impartial witness (by a person who is independent of the trial and cannot be unduly influenced by the people involved with the trial and who attends the informed consent process).
9. Negative pregnancy test for women of childbearing age.
10. Willingness to use reliable methods of contraception, and/or abstinence, for the duration of therapeutic product exposure.

Exclusion Criteria:

1. No evidence of clinical diagnosis of first-ever hemispheric ischemic stroke (codes ICD-10: I63.0 - I63.9).
2. Age <40 and > 80 years.
3. The National Institutes of Health Stroke Scale (NIHSS) score is <5 or >15 points.
4. Hemorrhagic stroke confirmed with CT/MRI.
5. Hemorrhagic transformation of ischemic stroke.
6. Recurrent ischemic stroke.
7. Parkinson's disease.
8. Epilepsy.
9. Demyelinating diseases of central nervous system.
10. Hereditary and degenerative diseases of the central nervous system.
11. Infectious diseases of central nervous system in medical history.
12. Traumatic brain injury with severe neurocognitive impairment in medical history.
13. Unstable angina pectoris.
14. The participant had a heart attack within 3 months prior to enrollment.
15. Heart failure class IV (NYHA).
16. 2nd and 3rd-degree atrioventricular block.
17. Systemic connective tissue disorders.
18. Chronic obstructive pulmonary disease (stage III or IV).
19. Acute surgical pathology
20. Severe decompensated heart failure/liver disease/kidney disease (including acute or chronic kidney/hepatic failure).
21. Medical history of oncology diseases, tuberculosis, immunodeficiency disorders, mental disorders or alcohol/drug addiction.
22. The investigator's decision not to enroll participant due to any severe condition that can be issue of safety or treatment efficacy.
23. Acute infectious diseases (influenza, SARS, etc.) within 4 weeks prior to enrollment.
24. Evidence of lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
25. Pregnancy or breastfeeding.
26. Any reason (including mental or physical states) that can affect participant's capability to follow protocol procedures.
27. The participant (or their relative) is affiliated with the clinical site or Sponsor company.
28. Participation in another clinical trial within 3 months prior to enrollment.
29. Evidence of hypersensitivity reactions or intolerance associated with ethylmethylhydroxypyridine, succinate drugs or Vitamin B6.
30. Medical contraindications for Mexidol®.
31. The written informed consent form (ICF) is not signed and personally dated by the participant or by an impartial witness.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Tatarstan Republican Clinical Hospital, Kazan'
  - Interregional Clinical Diagnostic Center, Kazan'
  - Kazan Clinical Hospital № 7, Kazan'
  - Research Institute of Experimental and Clinical Medicine, Novosibirsk
  - St. Petersburg Clinical Hospital № 26, Saint Petersburg
  - St. Petersburg Clinical Hospital № 2, Saint Petersburg
  - St. Petersburg "Nikolaevskaya" Hospital, Saint Petersburg
  - Samara Regional Clinical Hospital n.a. V. D. Seredavin, Samara
  - Samara Clinical Hospital № 1 n.a. N. I. Pirogov, Samara
  - City Hospital № 40 of Kurortny District, Sestroretsk
  - Vsevolozhsk Clinical Interdistrict Hospital, Vsevolozhsk

REFERENCES:
- [Result] Stakhovskaya LV, Shamalov NA, Khasanova DR, Melnikova EV, Agafiina AS, Golikov KV, Bogdanov EI, Yakupova AA, Roshkovskaya LV, Lukinykh LV, Lokshtanova TM, Poverennova IE, Shepankevich LA. [Results of a randomized double blind multicenter placebo-controlled, in parallel groups trial of the efficacy and safety of prolonged sequential therapy with mexidol in the acute and early recovery stages of hemispheric ischemic stroke (EPICA)]. Zh Nevrol Psikhiatr Im S S Korsakova. 2017;117(3. Vyp. 2):55-65. doi: 10.17116/jnevro20171173255-65. Russian. PMID 28665371
- [Result] Stakhovskaya LV, Mkhitaryan EA, Tkacheva ON, Ostroumova TM, Ostroumova OD. [Efficacy and safety of mexidol across age groups in the acute and early recovery stages of hemispheric ischemic stroke (results of additional sub-analysis of a randomized double blind multicenter placebo-controlled study, in parallel groups trial EPICA)]. Zh Nevrol Psikhiatr Im S S Korsakova. 2020;120(8. Vyp. 2):49-57. doi: 10.17116/jnevro202012008249. Russian. PMID 33016677
- See also: Results of a randomized double blind multicenter placebo-controlled, in parallel groups trial of the efficacy and safety of prolonged sequential therapy with mexidol in the acute and early recovery stages of hemispheric ischemic stroke (EPICA) — https://pubmed.ncbi.nlm.nih.gov/28665371/
- See also: Results of additional sub-analysis of a randomized double blind multicenter placebo-controlled study, in parallel groups trial EPICA — https://www.mediasphera.ru/issues/zhurnal-nevrologii-i-psikhiatrii-im-s-s-korsakova-2/2020/8-2/1199772982020082049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on protocol requirements at 11 clinical sites between March 2015 and May 2016. The first participant was enrolled on 6 March, 2015 and the last participant was enrolled on 20 February, 2016.
Pre-assignment Details: Of 151 screened participants, 150 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Mexidol® | Placebo
Started (The amount of participants that were randomized (ITT-population).) | 75 | 75
Completed (The amount of participants that completed the study and were included in PP-population.) | 61 | 63
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Population: ITT-population was used for description of baseline measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mexidol® | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 46 | 81
  >=65 years | 40 | 29 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.893 (10.246) | 61.52 (8.664) | 62.70 (9.53)
Age, Customized [Count of Participants; unit: Participants]
  Age, sub-groups: < 60 years | 27 | 32 | 59
  Age, sub-groups: 60-75 years | 36 | 40 | 76
  Age, sub-groups: 76-90 years | 12 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 31 | 31 | 62
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of the 6-point Modified Rankin Scale (mRS) at Visit 5 After Completion of the Course of Therapy for Both Arms
Description: The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke. Possible scores range from 0 (no symptoms at all) to 6 (dead) [6 point scale: min value 0, max value 6, higher scores mean a worse outcome].
Time Frame: Visit 5 (67-71 Day).
Population: Per Protocol Population (all participant assigned to Mexidol or Placebo) for calculating the mean score of the 6-point Modified Rankin Scale (mRS) at Visit 5 after completion of the course of therapy for both arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 61 | 63
score on a scale | 1.098 (0.768) | 1.46 (0.947)

2. Secondary Outcome: Mean Score of the 15-item The National Institutes of Health Stroke Scale (NIHSS) at Visit 5 After Completion of the Course of Therapy for Both Arms
Description: The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The individual scores from each item are summed in order to calculate a patient's total NIHSS score.
  The maximum possible score is 42 (severe stroke), with the minimum score being a 0 (no stroke symptoms).
Time Frame: Visit 5 (67-71 Day)
Population: Per Protocol Population (all participant assigned to Mexidol or Placebo) for calculating the mean score of the 15-item The National Institutes of Health Stroke Scale (NIHSS) at Visit 5 after completion of the course of therapy for both arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo (Group 2): Participants received Mexidol Placebo matching Mexidol solution IV 500 mg daily for 10 days, then Mexidol 125 mg orally 1 tablet 3 times a day for 8 weeks.
Arm/Group | Mexidol® | Placebo (Group 2)
Number analyzed (Participants) | 61 | 63
score on a scale | 1.689 (1.397) | 2.222 (1.442)

3. Secondary Outcome: Mean Score of the 10-item Barthel Index (BI) at Visit 5 After Completion of the Course of Therapy for Both Arms
Description: The Barthel Index (BI) is a prominent measure that assesses an individual's ability to perform activities of daily living (ADL) independently, reflecting their mobility and functional capacity. BI evaluates ten specific activities: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation, and stair climbing. Each activity is weighted based on the level of assistance required, with scores assigned as follows: 10 (independent), 5 (some assistance), and 0 (dependent).
  The BI's scoring system favors mobility and continence, resulting in a total score ranging from 0 to 100, where a higher score indicates greater functional independence. The index is widely utilized for assessing functional disability, particularly in rehabilitation settings for stroke patients and individuals with neuromuscular or musculoskeletal disorders, as well as in oncology care.
Time Frame: Time frame: Visit 5 (67-71 Day)
Population: Per Protocol Population (all participant assigned to Mexidol or Placebo) for calculating the mean score of the 10-item Barthel Index (BI) at Visit 5 after completion of the course of therapy for both arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 61 | 63
score on a scale | 96.066 (7.806) | 93.571 (12.229)

4. Secondary Outcome: Mean Score of the 21-item Beck Depression Inventory (BDI) at Visit 5 After Completion of the Course of Therapy for Both Arms.
Description: The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each item is scored 0 to 3 points for a total score range of 0 to 63. This range includes interpretation from 0-9 points (as normal condition) to over 30 points (as severe depression).
Time Frame: Visit 5 (67-71 Day)
Population: Per Protocol Population (all participant assigned to Mexidol or Placebo) for calculating the mean score of the 21-item Beck Depression Inventory (BDI) at Visit 5 after completion of the course of therapy for both arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 61 | 63
score on a scale | 2.213 (2.491) | 2.190 (2.693)

5. Secondary Outcome: Mean Score of on the EQ-5D-3L PRO Measure (VAS) at Visit 5 After Completion of the Course of Therapy for Both Arms.
Description: EQ-5D-3L is a concise, generic patient-reported outcome (PRO) measure of health consisting of five dimensions of health status (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (VAS). In the study version was used EQ-5D-3L that contains 3 severity levels for each dimension. The EQ VAS records the participants's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' (maximum indicated as 100 scores on VAS) and 'The worst health you can imagine' (minimum indicated as 0 on VAS).
Time Frame: Visit 5 (67-71 Day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 61 | 63
score on a scale | 83.82 (15.499) | 78.175 (17.52)

ADVERSE EVENTS:
Time Frame: Not less than 71 days for each participant
Description: Safety analysis was performed using ITT-population data (for 150 participants).
Arm/Group | Mexidol® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/75 | 3/75
Other Adverse Events (participants affected / at risk) | 21/75 | 16/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexidol® (N=75) | Placebo (N=75)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) — Severe recurrent IS
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) — Severe hemorrhagic stroke
Cholecystitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) — Acute cholecystitis
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexidol® (N=75) | Placebo (N=75)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatic enzyme increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Vascular disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days